CLINICAL TRIAL: NCT06093373
Title: Feasibility Study to Evaluate a New Hands-free Doppler Heart Rate Monitor Normally Used to Measure the Fetal Heart Rate
Brief Title: The Doppler Feasibility Study
Status: Completed | Type: Observational
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Other Study IDs: SCH-2798
Record Dates: First submitted 2023-09-25; First posted 2023-10-23 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-09

CONDITIONS: Heart Rate Measurements

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Comparison

SUMMARY:
The study is an exploratory research study looking at the feasibility, acceptability and accuracy of a doppler device compared with the gold standard ECG. It will take place in the sleep unit at Sheffield Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been referred for a cardio-respiratory polygraphy sleep study.
* Patients aged one month up to one year old.

Exclusion Criteria:

* Subjects whose parents/legal guardians/carers are not fluent in English, or who have special communication needs.
* Child anticipated to become distressed with additional sensor.
* Child too clinically unwell to take part (as decided by clinical staff).

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 1-12 months admitted to the Sleep Unit at Sheffield Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
The accuracy of the system in 15 patients, when compared with the gold standard ECG | 1 hour
The acceptability of the sensor to the child as viewed by the parent | 1 hour
  As measured by researcher designed questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, Sheffield Children's Hospital, Sheffield, United Kingdom